CLINICAL TRIAL: NCT04053881
Title: A Multicenter, Noninterventional, Prospective Study to Assess the Effectiveness of Certolizumab Pegol in Patients With Moderate to Severe Plaque Psoriasis in Daily Practice
Brief Title: A Study to Assess How Well Certolizumab Pegol Works in Patients With Moderate to Severe Plaque Psoriasis as Part of Routine Clinical Practice
Acronym: CIMREAL
Status: Completed | Type: Observational
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: PS0026
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis; Cimzia; Certolizumab pegol
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Certolizumab pegol: Plaque psoriasis patients who have been newly prescribed certolizumab pegol (CZP).
  Interventions: Drug: Certolizumab pegol

INTERVENTIONS:
Drug: Certolizumab pegol — Active Substance: Certolizumab Pegol Pharmaceutical Form: Prefilled syringe Concentration: 200 mg/ml Route of Administration: Subcutaneous injection
  Other Names: Cimzia; CDP870

SUMMARY:
The purpose of the study is to assess the effectiveness of certolizumab pegol in patients with moderate to severe plaque psoriasis as part of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥18 years of age at observational point 1
* The patient must have a clinical diagnosis of moderate to severe Plaque psoriasis according to the diagnostic criteria used by the physician in routine clinical practice
* The patient has an available PASI assessment prior to the first certolizumab pegol dose according to the standard of care
* The patient must be newly prescribed with certolizumab pegol
* If a patient is participating in an ongoing investigational study, then he/she will not be able to take part in this study

Exclusion Criteria:

Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Plaque psoriasis patients who have been newly prescribed certolizumab pegol (CZP).
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving Psoriasis Area Severity Index 75% response at observational point 2 | From Baseline up to Week 21
  The Psoriasis Area Severity Index (PASI75) response assessments are based on at least 75 % improvement in the PASI score from Baseline. The PASI score is a measure of the average redness, thickness, and scaliness of the psoriatic skin lesions with a score of 0 (clear) to 4 (very marked).

SECONDARY OUTCOMES:
Change from Baseline in Dermatology Life Quality Index score at observational point 2 | From Baseline up to Week 21
  The Dermatology Life Quality Index (DLQI) consists of questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. The DLQI score ranges from 0 to 30 with higher scores indicating lower health-related quality of life (HRQoL).
Change from Baseline in Dermatology Life Quality Index score at observational point 4 | From Baseline up to Week 56
  The Dermatology Life Quality Index (DLQI) consists of questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. The DLQI score ranges from 0 to 30 with higher scores indicating lower health-related quality of life (HRQoL).
Percentage of patients achieving Psoriasis Area Severity Index 75% response at observational point 4 | From Baseline up to Week 56
  The Psoriasis Area Severity Index (PASI75) response assessments are based on at least 75 % improvement in the PASI score from Baseline. The PASI score is a measure of the average redness, thickness, and scaliness of the psoriatic skin lesions with a score of 0 (clear) to 4 (very marked).
Percentage of patients achieving Psoriasis Area Severity Index 90% response at observational point 2 | From Baseline up to Week 21
  The Psoriasis Area Severity Index (PASI90) response assessments are based on at least 90 % improvement in the PASI score from Baseline. The PASI score is a measure of the average redness, thickness, and scaliness of the psoriatic skin lesions with a score of 0 (clear) to 4 (very marked).
Percentage of patients achieving Psoriasis Area Severity Index 90% response at observational point 4 | From Baseline up to Week 56
  The Psoriasis Area Severity Index (PASI90) response assessments are based on at least 90 % improvement in the PASI score from Baseline. The PASI score is a measure of the average redness, thickness, and scaliness of the psoriatic skin lesions with a score of 0 (clear) to 4 (very marked).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (79):
- Belgium (7):
  - Ps0026 101, Brussels
  - Ps0026 103, Brussels
  - Ps0026 107, Brussels
  - Ps0026 102, Leuven
  - Ps0026 110, Maldegem
  - Ps0026 109, Mons
  - Ps0026 104, Namur
- Canada (8):
  - Ps0026 208, London
  - Ps0026 209, London
  - Ps0026 201, Markham
  - Ps0026 210, Newmarket
  - Ps0026 203, St. John's
  - Ps0026 212, Toronto
  - Ps0026 205, Waterloo
  - Ps0026 204, Winnipeg
- Czechia (3):
  - Ps0026 301, Prague
  - Ps0026 303, Prague
  - Ps0026 302, Uherské Hradiště
- France (5):
  - Ps0026 408, Amiens
  - Ps0026 404, Lorient
  - Ps0026 409, Poitiers
  - Ps0026 403, Rennes
  - Ps0026 407, Toulon
- Germany (18):
  - Ps0026 512, Bielefeld
  - Ps0026 532, Bogen
  - Ps0026 525, Dresden
  - Ps0026 506, Düren
  - Ps0026 521, Freiburg im Breisgau
  - Ps0026 529, Gladbeck
  - Ps0026 523, Hamburg
  - Ps0026 518, Karlsruhe
  - Ps0026 519, Leipzig
  - Ps0026 537, Magdeburg
  - Ps0026 530, Memmingen
  - Ps0026 516, Merzig
  - Ps0026 517, München
  - Ps0026 527, München
  - Ps0026 515, Nuremberg
  - Ps0026 501, Potsdam
  - Ps0026 511, Quedlinburg
  - Ps0026 505, Remscheid
- Greece (9):
  - Ps0026 603, Athens
  - Ps0026 609, Athens
  - Ps0026 610, Athens
  - Ps0026 601, Chaïdári
  - Ps0026 606, Larissa
  - Ps0026 608, Pátrai
  - Ps0026 607, Piraeus
  - Ps0026 604, Thessaloniki
  - Ps0026 605, Thessaloniki
- Italy (13):
  - Ps0026 707, Bari
  - Ps0026 714, Bologna
  - Ps0026 711, Brescia
  - Ps0026 712, Catania
  - Ps0026 710, Florence
  - Ps0026 702, Genova
  - Ps0026 706, L’Aquila
  - Ps0026 701, Napoli
  - Ps0026 709, Roma
  - Ps0026 713, Roma
  - Ps0026 704, San Donato Milanese
  - Ps0026 715, Torino
  - Ps0026 708, Torrette DI Ancona
- Spain (6):
  - Ps0026 807, Badalona
  - Ps0026 809, Barcelona
  - Ps0026 812, Barcelona
  - Ps0026 804, Pontevedra
  - Ps0026 806, Sant Joan Despí
  - Ps0026 818, Vigo
- United Kingdom (10):
  - Ps0026 902, Bradford
  - Ps0026 909, Dunfermline
  - Ps0026 914, Glasgow
  - Ps0026 916, Hertfordshire
  - Ps0026 911, Kingston upon Thames
  - Ps0026 905, Leeds
  - Ps0026 904, Newcastle upon Tyne
  - Ps0026 901, Salford
  - Ps0026 915, Wakefield
  - Ps0026 908, York

IPD SHARING:
Plan to Share IPD: No
Data from non-interventional studies is outside of UCB's data sharing policy and is unavailable for sharing.

REFERENCES:
- [Derived] Korge B, Vanhooteghem O, Lynde CW, Machovcova A, Perrussel M, Lazaridou E, Marasca C, Sarro DV, Pousa ID, Fierens F, Williams P, Shimizu S, Heidbrede T, Warren RB. Certolizumab Pegol for the Treatment of Plaque Psoriasis in Routine Clinical Practice: One-Year Results from the CIMREAL Study. Dermatol Ther (Heidelb). 2024 Aug;14(8):2077-2092. doi: 10.1007/s13555-024-01210-3. Epub 2024 Jun 27. PMID 38937404